CLINICAL TRIAL: NCT04878146
Title: Comparaison Entre la Sacrocervicopexie (SCP) et la Fixation Sacro-spinale (FSS) du Col utérin Dans le Traitement du Prolapsus génital: Etude Prospective randomisée: Etude "ProSac "
Brief Title: Sacrocolpopexy Versus Sacro-spinous Fixation for Prolapse Treatment
Acronym: ProSac
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Chahin Achtari, Dr, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUV
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacrocolpopexy (Active Comparator): Used as the standard intervention for prolapse
  Interventions: Procedure: Subtotal hysterectomy; Procedure: Sacrocolpopexy
- Sacro-spinous fixation (Experimental): To be demonstrated as non inferior
  Interventions: Procedure: Sacro-spinous fixation; Procedure: Subtotal hysterectomy

INTERVENTIONS:
Procedure: Sacro-spinous fixation — Uterine cervix will be attached to the sacro-spinous ligament
  Other Names: Richter operation
  Arms: Sacro-spinous fixation
Procedure: Subtotal hysterectomy — Done on both arms
Procedure: Sacrocolpopexy — Uterine cervix is attached to sacral promontory with two synthetic meshes
  Arms: Sacrocolpopexy

SUMMARY:
Prolapse is a condition that causes up to 13% of women to have surgery in their lifetime. There are many surgical techniques for the treatment of prolapse, each with its advantages and disadvantages. The techniques by vaginal approach aim to put back in tension the supporting tissue, the endopelvic fascia, damaged and released. This technique has the advantage of not causing an abdominal scar, a quick recovery and often little pain. In contrast, the use of already damaged native tissue results in a recurrence rate of up to 15% to 30%.

The other technique is the abdominal route either by laparotomy or by a minimally invasive approach such as laparoscopy, assisted or not by robotics. With this technique, we use prosthetic material introduced around the vaginal wall without opening the latter, therefore without contamination and without dissection of the vaginal wall.

During upper surgery, a subtotal hysterectomy is performed, that is to say that the uterine cervix is preserved and serves as an anchoring point for the synthetic nets which are attached to the cervix and then sutured to the promontory of the sacrum. (sacrocervicopexy).

In the vaginal route, a total hysterectomy is traditionally performed and the vaginal dome is sutured to the sacro-spinal ligament (Richter's operation). The stitches are then passed through the thickness of the often thin vaginal wall constituting a possible release point of the assembly. There are currently no studies that compare prosthetic sacrocervicopexy with fixation of the remaining cervix to the sacro-spinal ligament without prosthesis, and repair of the endopelvic fascia with native tissue. The study consists of performing a subtotal hysterectomy by minimally invasive approach in both cases and then randomize for either a prosthetic sacrocervicopexy or fixation of the remaining cervix to the sacro-spinal ligament via the abdominal or vaginal route.

DETAILED DESCRIPTION:
Genital prolapse is caused by the collapse of the supporting structures of the pelvic organs. This results in the organs sliding down through the pelvic hiatus. The pelvic organs involved are the bladder, which rests on the anterior vaginal wall like a hammock made of supportive connective tissue called the anterior endopelvic fascia. When too much stress is placed on this support tissue, microtrauma or tears gradually weaken this tissue, which relaxes and causes the bladder to gradually lower. In the same way, the rectum is separated from the posterior vaginal wall by this same endopelvic fascia which can suffer the same kind of lesion with the same consequences. The middle compartment, i.e. the top of the vagina is made up of the cervix which is supported by a condensation of this endopelvic tissue in the form of ligaments that suspend this cervix in the center of the pelvic cavity. If these ligaments weaken, the uterus, or the "vaginal cuff" in the event of a previous hysterectomy, will also gradually lower, or even externalize. The middle compartment is considered the keystone of pelvic organ support. All interventions to correct severe prolapse should include suspension of the middle compartment. Traditionally, the sacro-spinal ligament is used during the intervention via the low approach and the sacral promontory via the high approach.

There is a classification (Pelvic Organ Prolapse Quantification or POP-Q) in stages of descent of the pelvic organs. At the first stage, the organs are not exteriorized and in most cases asymptomatic. In the second stage, the vaginal walls reach the vaginal introitus and begin to cause symptoms such as pelvic discomfort or heaviness, whether or not associated with functional disorders of the organs involved. In the following stages, the patients are generally symptomatic.

Prolapse is a condition that causes up to 13% of women to have to have surgery in their lifetime. It causes both an impairment of the quality of life by the discomfort caused by the externalization of the organs and by the functional disorders that it causes, such as urinary or fecal incontinence, bladder emptying disorder, sexual disorders, etc. all of these disorders can be measured by dedicated questionnaires and validated in this population.

There are many surgical techniques for the treatment of prolapse, each with its advantages and disadvantages. The techniques by vaginal approach aim to put back in tension of the native supporting tissue damaged and released. This technique has the advantage of not causing an abdominal scar, a quick recovery and often little pain. On the other hand, the use of already damaged tissue results in a recurrence rate of up to 15-30%. In an attempt to reduce this rate of recurrence, by taking the example of abdominal hernia surgery, prosthetic reinforcements have started to be used in order to make the repair more solid and durable. The prostheses were introduced through a vaginal incision (naturally contaminated medium) and directly under the mucosa. It turned out that a reduction in recurrence was achieved, especially in the anterior compartment, but at the cost of complications directly linked to the use of prostheses such as erosions of the vaginal mucosa, infections and, when using implantation kits supplied by industry, pain that is often difficult to treat.

The other technique is the abdominal route either by laparotomy or by a minimally invasive approach such as laparoscopy, assisted or not by robotics. With this technique, prosthetic material is also used but it is introduced around the vaginal wall without opening it, therefore without contamination and without dissection of the vaginal wall, with a much lower rate of erosion or other complication.

Many studies have compared these different techniques without reaching a definitive conclusion on the best approach. The use of synthetic material introduced vaginally using kits has recently been the subject of warnings from the FDA due to the sometimes severe complications followed by a gradual withdrawal of these products or even a ban in most Anglo-Saxon countries. On the other hand, the use by the abdominal route not causing the same complications has not been questioned by the FDA

. In our department, the management of symptomatic prolapse involves two techniques, vaginal without prosthesis or minimally invasive abdominal with prosthesis, according to various criteria such as age, surgical history or severity of the prolapse. During upper surgery, a subtotal hysterectomy is performed, i.e. the uterine cervix is preserved and serves as an anchoring point for the synthetic nets which are attached to the cervix and then sutured to the promontory of the sacrum. (sacro-cervicopexy). In the vaginal route, a total hysterectomy is traditionally performed and the vaginal dome is sutured to the sacro-spinal ligament (Richter's operation). The stitches are then passed through the thickness of the often thin vaginal wall constituting a possible release point of the assembly. There are currently no studies that compare prosthetic sacro-cervicopexy with fixation of the remaining cervix to the sacro-spinal ligament without prosthesis and repair of the endopelvic fascia with native tissue. The study consists of performing a subtotal hysterectomy by minimally invasive first in both cases and then randomise for the mode of suspension of the uterine cervix, either a prosthetic sacro-cervicopexy or to fix the remaining cervix to the sacro-sinous ligament by abdominal or vaginal route. We would thus obtain more solid anchoring points at the level of the middle compartment with less risk of dropping and a more lasting result.

The main objective is to demonstrate that this new intervention gives similar results to the reference intervention by the upper route. For this we use a composite definition of the success of the intervention which takes into account the anamnestic aspect, the absence of a sensation of prolapse, the clinical examination, the absence of measurable prolapse, and the absence of secondary surgery. The secondary objectives are to ensure a similar improvement in the quality of life in the two groups by relying on specific questionnaires validated for this indication.

ELIGIBILITY:
Inclusion Criteria:

Patients who:

1. Have symptomatic prolapse, degree ≥ 2
2. Want surgical management
3. Accept subtotal hysterectomy
4. Accept the idea of being in the arm of the study, which involves the placement of prosthetic material
5. After explaining and reading the information sheet, have understood and signed the consent form

Exclusion Criteria:

1. Refuse hysterectomy
2. Refuse the idea of having prosthetic material implanted
3. Prefer conservative management
4. Have insufficient understanding of French
5. Still wish a pregnancy
6. Are not in a condition to withstand surgery of this type

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Non inferiority of sacro-spinous fixation compared to sacrocolpopexy after 1 year | 1 year
  Anatomical and symptomatic definition of success measured by validated questionnaires

SECONDARY OUTCOMES:
Operative time | Immediately after operation
  Measure of operative time
Complications | 30 days
  Measured with Clavien Dindo classification

IPD SHARING:
Plan to Share IPD: No